CLINICAL TRIAL: NCT02511613
Title: A Study of Safety, Functional and Anatomical Effect of Squalamine Lactate Ophthalmic Solution, 0.2% Administered Twice Daily in Subjects With Neovascular Age-related Macular Degeneration
Brief Title: Effect of Squalamine Lactate Ophthalmic Solution, 0.2% in Subjects With Neovascular Age-Related Macular Degeneration
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Company decision
Sponsor: Ohr Pharmaceutical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OHR-1501
Record Dates: First submitted 2015-07-27; First posted 2015-07-30 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — squalamine; Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Monthly intravitreal ranibizumab plus Placebo Ophthalmic solution
  Interventions: Drug: Placebo Ophthalmic Solution; Drug: ranibizumab
- Active (Active Comparator): Monthly intravitreal ranibizumab plus Squalamine Lactate Ophthalmic solution 0.2%
  Interventions: Drug: Squalamine Lactate Ophthalmic Solution, 0.2%; Drug: ranibizumab

INTERVENTIONS:
Drug: Squalamine Lactate Ophthalmic Solution, 0.2% — Squalamine Lactate Ophthalmic Solution, 0.2% administered BID
  Other Names: Squalamine
  Arms: Active
Drug: Placebo Ophthalmic Solution — Placebo Ophthalmic Solution, administered BID
  Other Names: Placebo
  Arms: Placebo
Drug: ranibizumab — ranibizumab intravitreal injection
  Other Names: Lucentis®

SUMMARY:
The purpose of this study is to evaluate anatomical and functional effect of combination therapy of Squalamine Lactate Ophthalmic Solution, 0.2% administered twice daily with monthly ranibizumab intravitreal injections in patients with choroidal neovascularization due to AMD.

DETAILED DESCRIPTION:
Subjects with age-related macular degeneration who meet inclusion and exclusion criteria will be randomized to receive monthly intravitreal injections of ranibizumab (Lucentis®) with either Squalamine Lactate Ophthalmic solution 0.2% or placebo eye drops twice a day for 6 months. Subjects will be evaluated with clinical and imaging techniques.

ELIGIBILITY:
Inclusion Criteria:

* 50 years of age or older
* A diagnosis of choroidal neovascularization secondary to age-related macular degeneration (AMD) with choroidal neovascularization (CNV) comprising at least 50% of the total lesion area in the study eye
* Central retinal thickness ≥ 300 μm and presence of subretinal fluid or cystoid edema by Optical Coherence Tomography (OCT)
* Best Corrected Visual Acuity (BCVA) of 20/40 to 20/320 by Early Treatment Diabetic Retinopathy Study (ETDRS) Protocol

Exclusion Criteria:

* Neovascularization secondary to any other condition than AMD in the study eye
* Blood occupying greater than 50% of the AMD lesion, or blood > 1.0 sq. mm underlying the fovea
* PED without associated subretinal fluid and/or cystic retinal changes
* Clinical evidence of diabetic retinopathy or diabetic macular edema in the study eye
* Confounding ocular conditions in the study eye which will affect interpretation of OCT, VA or assessment of macular appearance (e.g., cataract, epiretinal membrane, retinal vascular occlusive disease)
* Fibrosis or atrophy, retinal epithelial tear in the center of the fovea in the study eye or any condition preventing VA improvement
* Uncontrolled glaucoma in the study eye, or currently receiving topical glaucoma medication in the study eye

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-07; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Effect of combination therapy of ranibizumab monthly intravitreal injections with Squalamine Lactate Ophthalmic Solution, 0.2% on anatomy and function as assessed by retinal imaging and ETDRS BCVA in subjects with Age-Related Macular Degeneration | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Avner Ingerman, MD, Study Director — Ohr Pharmaceutical
Locations (4):
- United States (4):
  - Investigational Site, Beverly Hills, California
  - Investigational Site, Hagerstown, Maryland
  - Investigational Site, New York, New York
  - Investigational Site, Houston, Texas